CLINICAL TRIAL: NCT06657287
Title: Relationship Between Insulin Levels and Postprandial Hypotension in the Standard Mixed Meal Test in Adults
Brief Title: Postprandial Hypotension and Insulin Levels
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Rahime Evra KARAKAYA, Principal Investigator, Ankara Yildirim Beyazıt University
Other Study IDs: AnkaraYBU-KARAKAYA004
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Postprandial Hypotension; Hypoglycemia
Keywords: Hypotension; hypoglycemia; insulin; mixed meal; adults; postprandial
MeSH Terms: conditions — Hypoglycemia; Hypotension; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy adults: Adults with postprandial symptoms
  Interventions: Other: Mixed meal test

INTERVENTIONS:
Other: Mixed meal test — The biochemical parameters, blood pressure, and heart rates of participants undergoing the mixed meal test will be recorded over a 5-hour period.

SUMMARY:
The goal of this observational study is to learn about the relationship between postprandial hypotension and insulin levels in adults. The main question it aims to answer is:

Is the incidence of postprandial hypotension high in patients who undergo mixed meal test?

Is insulin level higher in individuals with postprandial hypotension compared to those without during a mixed meal test?

Patients with postprandial symptoms were scheduled for a mixed meal test, during which plasma glucose, insulin, C-peptide, blood pressure, and heart rate were measured at specific time points.

ELIGIBILITY:
Inclusion Criteria:

* Adults with postprandial symptoms

Exclusion Criteria:

* Individuals with prediabetes or diabetes,
* Those aged 65 and above,
* Patients using antihypertensive medications or with known hypertension,
* Those with active infections,
* Congestive heart failure,
* Peripheral artery disease,
* Advanced-stage dementia,
* Individuals who could not provide a history or were unable to cooperate,
* Patients using medications that could induce hypoglycemia (oral antidiabetics, insulin, beta-blockers, hydroxychloroquine, bromocriptine, etc.)
* Those with conditions that could cause hypoglycemia (uncontrolled hypothyroidism, adrenal insufficiency, growth hormone deficiency, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who apply to the Endocrinology Clinic of Ankara Bilkent City Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | During mixed meal test (baseline, 30., 60., 90., 120., 180., 240., 300. min)
  mmHg
Blood glucose | During mixed meal test (baseline, 30., 60., 90., 120., 180., 240., 300. min)
  mg/dL
Blood insulin | During mixed meal test (baseline, 30., 60., 90., 120., 180., 240., 300. min)
  uIU/mL

SECONDARY OUTCOMES:
Blood C-peptide | During mixed meal test (baseline, 30., 60., 90., 120., 180., 240., 300. min)
  ng/mL
Diastolic blood pressure | During mixed meal test (baseline, 30., 60., 90., 120., 180., 240., 300. min)
  mmHg
Heart rate | During mixed meal test (baseline, 30., 60., 90., 120., 180., 240., 300. min)
  bpm

CONTACTS AND LOCATIONS:
Overall Officials: Rahime E Karakaya, PhD, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No